CLINICAL TRIAL: NCT04088955
Title: A Pragmatic, Non-Interventional Study of DigiMeds™ in Combination With Standard of Care for Treatment of Patients With Cancer
Brief Title: A Digimed Oncology PharmacoTherapy Registry
Acronym: ADOPTR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Proteus Digital Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO 1676
Record Dates: First submitted 2019-09-10; First posted 2019-09-13 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2019-09

CONDITIONS: Colon Cancer; Breast Cancer; Rectal Cancer
Keywords: DigiMeds; Capecitabine; Standard of Care
MeSH Terms: conditions — Colonic Neoplasms; Breast Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: DigiMeds — Digitized Capecitabine

SUMMARY:
DigiMeds™ are medications with FDA-approved ingestible sensors (IS), a wearable sensor patch (patch), and a mobile app, which records time-stamped medication type and dose alongside biometric activity.

The aim of this registry is to collect and analyze data on the use of DigiMeds™ and a digital feedback system on medication adherence, patient-provider communication, and data-driven optimization of therapy for cancer patients.

DETAILED DESCRIPTION:
Patients will be prescribed the DMP and DigiMeds™ (capecitabine or supportive medications) by their healthcare provider. The pharmacy will co-encapsulate the prescribed medication with a sensor.

The actual doses of DigiMeds™ will be based on standard of care as prescribed by treating physician. Patients will be instructed in the use of the DigiMeds™ and the DMP based on standard of care plus use of the DMP system.

Every effort should be made to take the DigiMeds™ as prescribed.

Patients in this study will be given the option to use their personal smartphone or will be provided a provisioned iPad to use for the duration of the study. Each patient will receive a Starter Kit comprised of two wearable sensor pods, adhesive strips, and instructions. Additionally, some kits may contain the provisional iPad Mini and charger for those without an approved smart device. Should a device malfunction occur, such as a broken pod, the patient can replace it with their spare pod. Broken pods should be returned to Proteus as soon as possible and all pods must be returned to the clinic upon completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Prescribed treatment with DigiMeds™
* Have an Android or iOS-enabled device (e.g., iPhone, iPad, Samsung) or be willing to use a Proteus issued iOS device
* Signed consent form

Exclusion Criteria:

* Receiving palliative or hospice care services (i.e., proxy for <12 months life expectancy)
* Not proficient in the English language
* Have impaired cognitive ability
* For women: current pregnancy
* Have skin sensitivity to adhesives or active/chronic dermatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with colon, rectal, or breast cancer and diagnosed therapy with capecitabine.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-09-06 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Compare the duration of actual vs. intended treatment for cancer patients on capecitabine who are prescribed capecitabine with sensor. | Up to 6 months from the date of inclusion into study
  Determine how long patients can stay on treatment when using DigiMeds

CONTACTS AND LOCATIONS:
Overall Officials: Sinette Heys, Study Director — Proteus Digital Health
Locations (1):
- Carolina Blood and Cancer Care, Rock Hill, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No